CLINICAL TRIAL: NCT02967562
Title: Comparison of a Sustained Inflation to Shorter Inflation Breaths During Resuscitation at Delivery of Prematurely Born Infants
Brief Title: Neonatal Resuscitation - Sustained Inflations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCH16-155
Record Dates: First submitted 2016-11-15; First posted 2016-11-18 (Estimated); Results first posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2018-03

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inflation Breaths (Active Comparator): Five 'inflation breaths' lasting two - three seconds
  Interventions: Other: Inflation Breaths
- Sustained inflation (Experimental): One fifteen second 'sustained inflation'
  Interventions: Other: Sustained Inflation

INTERVENTIONS:
Other: Inflation Breaths
  Arms: Inflation Breaths
Other: Sustained Inflation
  Arms: Sustained inflation

SUMMARY:
This study compares a fifteen second sustained inflation (SI) to five repeated two - three second 'inflation breaths' during resuscitation at delivery of infants born prematurely.

DETAILED DESCRIPTION:
Around 10% of newborns will require some form of assistance after delivery, with babies born more prematurely more likely to require resuscitation

Current UK guidelines advise initial resuscitation with the delivery of five 'inflation breaths' lasting 2-3 seconds with peak inflation pressure of 30cmH2O (20-25cm H2O in premature neonates). Previous studies have shown that despite resuscitation training, clinicians in both simulated and real resuscitation scenarios do not deliver the recommended duration of inflation breaths. This, combined with leaks around the facemask often being as large as 50% or greater, contributes to low expired tidal volumes during resuscitation, thus increasing the likelihood of hypoxia and delay in establishing effective respiration.

The use of sustained inflations (up to 15 seconds), rather than intermittent shorter inflation breaths, has shown promising results, with reduction in the need for intubation, and the need for and duration of mechanical ventilation. Around 30% of units in Germany use sustained inflations as first line delivery room management, as do many other hospitals around the world. Resuscitation guidelines from the USA, UK and Europe suggest that sustained inflations should be researched further.

Several studies have shown that for several lengths of inflation breaths, the expired tidal volume achieved is higher if the baby makes respiratory effort during the inflation (active inflation) and that stimulation of spontaneous respiratory effort is a key part in establishing an FRC, enabling spontaneous breathing, and increasing the likelihood of successful resuscitation.

To date, there are no studies directly comparing whether prolonged inflations are more successful at provoking an inspiration than other methods of resuscitation. We therefore aim to compare a 15 second sustained inflation to repeated shorter inflations to determine which is more effective.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at less than 34 weeks gestation requiring resuscitation at delivery

Exclusion Criteria:

* Major congenital abnormalities
* Parents have previously expressed lack of consent for study

Ages: 0 Minutes to 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2016-11; Primary Completion 2018-03 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Greenough, MD, FRCPCH, Study Director — King's College London
Locations (1):
- King's College Hospital, London, United Kingdom

REFERENCES:
- [Derived] Hunt KA, Ali K, Dassios T, Milner AD, Greenough A. Sustained inflations versus UK standard inflations during initial resuscitation of prematurely born infants in the delivery room: a study protocol for a randomised controlled trial. Trials. 2017 Nov 28;18(1):569. doi: 10.1186/s13063-017-2311-y. PMID 29179773

RESULTS

PARTICIPANT FLOW:
Groups:
- Inflation Breaths: Five 'inflation breaths' lasting two - three seconds
  Inflation Breaths
- Sustained Inflation: One fifteen second 'sustained inflation'
  Sustained Inflation
Period: Overall Study
Arm/Group | Inflation Breaths | Sustained Inflation
Started | 32 | 31
Completed | 30 | 30
Not Completed | 2 | 1
Not completed — Consent not obtained | 1 | 0
Not completed — High leak precluding analysis | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inflation Breaths | Sustained Inflation | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Full Range); unit: post menstrual weeks] | 29.7 [23.1 to 33.6] | 30.6 [24 to 33.7] | 30.3 [23.3 to 33.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 14 | 20 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Expiratory Tidal Volume
Description: Expiratory tidal volume during the first minute of resuscitation
Time Frame: one minute
Measure: Median (Full Range); unit: ml/kg/min
Arm/Group | Inflation Breaths | Sustained Inflation
Number analyzed (Participants) | 30 | 30
ml/kg/min | 153 [18 to 385] | 194 [45 to 505]

2. Secondary Outcome: End Tidal Carbon Dioxide Level
Description: end tidal carbon dioxide level during resuscitation
Time Frame: 10 minutes
Measure: Median (Full Range); unit: mmHg
Arm/Group | Inflation Breaths | Sustained Inflation
Number analyzed (Participants) | 30 | 30
mmHg | 28.6 [1.9 to 46] | 34.2 [1.4 to 80.5]

3. Other Pre Specified Outcome: Mechanical Ventilation
Description: Duration of mechanical ventilation ini first 48 hours
Time Frame: 48 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Inflation Breaths | Sustained Inflation
Number analyzed (Participants) | 30 | 30
hours | 32.5 [0 to 48] | 17 [0 to 48]

4. Other Pre Specified Outcome: Adverse Effects
Description: Rates of intraventricular haemorrhage, significant patent ductus arteriosus, and pneumothorax
Time Frame: First week of life
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Until study completion, maximum of 6 months.
Arm/Group | Inflation Breaths | Sustained Inflation
All-Cause Mortality (participants affected / at risk) | 3/32 | 2/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT02967562/Prot_SAP_000.pdf